CLINICAL TRIAL: NCT05967013
Title: Evaluation by Magnetic Resonance Imaging of Intramuscular Injections Performance in Thigh With 2 Configurations of the Needle-free Injector ZENEO®.
Acronym: MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Crossject (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CJTMRIZ2101
Record Dates: First submitted 2023-07-20; First posted 2023-08-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Needle-free Injector
Keywords: Needle-free injector; Magnetic Resonance Imaging; Intramuscular; Injection
MeSH Terms: interventions — Injections

STUDY DESIGN:
Intervention Model Description: An open-label single-dose, 4-period cross-over, randomized, non-comparative mono-centric study where 0.625 mL of a saline solution will be injected in the thigh (on bare skin or through clothing) with the ZENEO® injector to healthy subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4-period cross-over (Experimental): After a screening period of a maximum of 21 days, eligible subjects will be randomized in a 1:1:1:1 allocation ratio to one of the 4 treatment sequences (settings):
  * Sequence 1: A&B in Period 1 / C&D in Period 2
  * Sequence 2: D&A in Period 1 / B&C in Period 2
  * Sequence 3: C&D in Period 1 / A&B in Period 2
  * Sequence 4: B&C in Period 1 / D&A in Period 2
  Setting definitions:
  * Setting B = volume "0.64mL" of physiological serum with ZENEO® injector, setting "GAMMA" - Bare skin.
  * Setting A = volume "0.64mL" of physiological serum with ZENEO® injector, setting "GAMMA" - Through Clothing.
  * Setting D = volume "0.64mL" of physiological serum with ZENEO® injector, setting "GAMMA low" - Bare skin.
  * Setting C = volume "0.64mL" of physiological serum with ZENEO® injector, setting "GAMMA low" - Through Clothing.
  Interventions: Combination Product: Injections in thigh of 0.625 mL of physiological serum with ZENEO® injector, on bare skin and through clothing.

INTERVENTIONS:
Combination Product: Injections in thigh of 0.625 mL of physiological serum with ZENEO® injector, on bare skin and through clothing. — All injections with ZENEO® injector will be performed in the thigh. Due to MRI performance constraints, injection sites will be identified on the same thigh/leg at each treatment period: first leg on treatment period 1, opposite leg on treatment period 2.
  At each treatment period, two injection sites will be identified spaced 8 to 15 cm apart. The 2 injections should be performed on the same leg at each treatment period.
  In total, 2 injections will be performed per treatment period, and subjects will receive 4 injections during the study :
  * 2 injections on bare skin: 1 with GAMMA configuration of ZENEO® injector & 1 with GAMMA-Low configuration ZENEO® injector.
  * 2 injections through clothing: 1 with GAMMA configuration of ZENEO® injector & 1 with GAMMA-Low configuration ZENEO® injector.

SUMMARY:
The aim of this study is to establish with measures of clinical parameters by Magnetic Resonance Imaging (MRI) (e.g. crossing of the muscle fascias, length of run, injection depth, volume injected) performance of 2 configurations of the needle-free injector when used for intramuscular injection on bare skin or through clothing.

DETAILED DESCRIPTION:
The development of needle-free injection devices has been motivated by a need for safer and more user-friendly injection devices that can prevent needle-stick injuries and contamination as well as improve patient comfort and treatment. As a growing number of drugs need to be injected or self-injected, needle-free devices are an attractive alternative to the conventional needle, especially in situation of emergency.

A medical emergency requires quick action to ward off a risk of imminent death and long-term sequelae, or to manage a situation of stress or crisis. Study's sponsor has developed an innovative, needle-free, prefilled, single use, disposable injector called ZENEO®. Unlike other needle-free injection devices, ZENEO® does not resemble a syringe in order to make injections with the device as natural and user friendly

The prefilled, single use, combined system of ZENEO® makes it ready to use for any type of drug or vaccine that needs to be injected into the skin (intradermal), under the skin (subcutaneous) or into the muscle (intramuscular).

According to regulatory requirements for market-authorization submission, proof of performance of ZENEO® injector for intramuscular (i.m.) injection must be established.

For each drug development as combination with the ZENEO® injector, clinical investigations will be conducted to study the relative bioavailability of the medicinal product when injected either with ZENEO® or with a conventional syringe.

Performance profile of ZENEO® injector for i.m. injection on the thigh with a target volume of 0.625 milliliter (mL) of an aqueous solution have been calculated and must be verified by clinical data in order to demonstrate successful delivery of the intended medication(s) to the target tissues, achieving therapeutic bioavailability, or reaching another appropriate endpoint in humans.

This is the reason why this clinical study CJTMRIZ2101 will be conducted.

After a screening period of a maximum of 21 days, eligible subjects will be randomized in a 1:1:1:1 allocation ratio and will receive 2 intramuscular injections on the thigh with ZENEO® pre-filled with 0.64 mL of physiological serum, at 2 treatments periods - Period 1 (P1) and Period 2 (P2) - separated by a wash-out period of at least 7 days. Each injection will be spaced of no more than 5 minutes. Within 10 minutes after the first injection and no more than 5 minutes after the second injection, subjects will be settled for the MRI sequences acquisition (about 20 minutes) so that the MRI acquisition should end no more than 30 minutes (+/- 5 minutes) after the first injection.

A follow-up visit (phone contact) will systematically be performed two days after Day 1 of P1 and Day 1 of P2, in order to confirm there is no safety concern on the injection site and to confirm the subject's well-being. If a subject indicates a pain score >5 or any significant anomaly an on-site follow-up visit will be organized within 7 days after each follow-up phone call.

A total of 50 healthy volunteers will be enrolled in this investigation with at least 30% of males and 30% of females are expected.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female volunteers aged between 18 and 59 years (inclusive) at the Screening Visit.
2. Female subjects of childbearing potential (i.e., fertile, following menarche and until becoming post-menopausal unless permanently sterile: neither post-menopausal nor surgically sterile) who are sexually active with a non-sterile male partner must be willing to use one of the following effective contraceptive methods throughout the study and for 30 days after the last study intervention:

   1. Combined estrogen and progestogen-containing or progestogen-only hormonal contraception associated with inhibition of ovulation, started at least 4 weeks prior to the first study intervention;
   2. Intrauterine device placed at least 4 weeks prior to the first study intervention, and condom for the male partner;
   3. Simultaneous use of a diaphragm or cervical cap with intravaginally applied spermicide and for the male partner a male condom;
   4. Sterile male partner (i.e. vasectomized since at least 6 months prior to the first study intervention);
   5. Sexual abstinence (when in line with the preferred and usual subject lifestyle). Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) is not acceptable.
3. Female subjects of non-childbearing potential must be:

   1. Post-menopausal female (absence of menses for 12 months prior to the first [if applicable] study intervention); or
   2. Surgically sterile female (documented hysterectomy, or bilateral oophorectomy or bilateral tubal ligation/occlusion) or bilateral tubal ligation at least 6 months prior to the first [if applicable] study intervention).
4. Subject with BMI between ≥ 16.0 and < 35.0 kg/m² at the Screening Visit.
5. Injection sites must be clear of tattoos, scars and moles.
6. Affiliated to or covered by the French social security system.
7. Signed written consent given for participation in the study.

Exclusion Criteria:

1. Known Contra-Indication to i.m. injection.
2. Treatment with platelet inhibiting drugs within one week before inclusion.
3. Treatment with anticoagulant within four weeks before inclusion.
4. Any Contra-indication to MRI (ex: metallic intra-corporeal devices, claustrophobia, tremor or abnormal movements whatever the origin is).
5. A major illness during the 3 months before the screening period, that may interfere with the evaluation, as judged by the investigator
6. Any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary neurologic, dermatologic, psychiatric, renal, and/or other major disease or malignancy, as judged by the Investigator.
7. Any clinically significant abnormality following the Investigator's review of the physical examination, ECG and clinical study protocol-defined clinical laboratory tests at screening or admission to the clinical unit.
8. A pulse < 45 or > 90 bpm; mean systolic blood pressure > 140 mmHg; mean diastolic blood pressure > 90 mmHg (measurements taken in triplicate after subject has been resting in supine position for 5 minutes.
9. Current alcohol use > 21 units of alcohol per week for males and > 14 units of alcohol per week for females.
10. Regular exposure to substances of abuse (other than alcohol) within the past year.
11. Positive urine screen for drugs of abuse and for alcohol breath test at screening and before the first study intervention (P1). In case of a positive result, urine screen for drugs may be repeated once at the discretion of the Investigator.
12. Donation or loss of blood equal to or exceeding 500 mL during the 8 weeks before the first use of the Investigational Medicinal Device.
13. History of hypersensitivity or allergy to any topical disinfectant.
14. Positive testing at screening for current infection Human Immunodeficiency Virus (HIV), Hepatitis B and/or Hepatitis C.
15. Breastfeeding woman.
16. Positive pregnancy test at screening (β-Human Chorionic Gonadotropin test) and Check-in (Day1-P1) (urine test).
17. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.
18. Participation in another interventional clinical trial within 3 months prior to screening.
19. In custody due to administrative or legal decision or under tutelage or being admitted in a sanitary or social institution.
20. Vulnerable subjects, e.g. persons in detention.
21. Subject is the Principal Investigator or any Sub-Investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the study or employee of the Sponsor (or representatives).

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
Intra-muscular injection success rate | Within 20 minutes after injection with the ZENEO® injector.
  The intra-muscular injection success rate defined as the muscle fascias are crossed by the saline solution as objectified by MRI:
  * Success of crossing the muscle fascia defined as injection 'depth in the muscle greater than 0 mm
  * Success of intra-muscular injection defined as injection 'depth in the muscle greater than 5 mm

SECONDARY OUTCOMES:
Injection parameters evaluated by MRI | Within 20 minutes after injection with the ZENEO® injector
  * Distance in millimeters (mm) :
    * Maximal vertical depth of the injection
    * Length of the injectate run
    * Width of the injectate in the muscle
    * Maximum vertical depth of the injectate in the muscle
    * Derma depth
    * Skin-to-muscle distance
    * Skin-to-bone distance
    * Subcutaneous tissue thickness
    * Fat thickness (when applicable)
  * Volume in milliliters (mL) :
    . Estimated volume of physiological serum injected into the muscles
  * Direction of injectate (head/Vertical/Foot)
  * Imaging gradation :
    * Image Quality (0 to 4)
    * Visibility of injectate (0 to 4)
Occurence of local tolerability events | At 5 minutes after each injection with the ZENEO® injector at Day 1 of each treatment period
  Any signs of erythema, swelling, bruising, allergic reaction and bleeding
Anthropometric characteristics of thighs (left and right) acquired by Ultrasound (no contrast agent will be used) | To be performed once during the study
  * Derma depth (mm)
  * Subcutaneous tissue depth (mm)
  * Skin-to-muscle distance (mm)
  * Skin-to-bone distance (mm)
  * Fat thickness (when applicable(mm)
Average pain rating | At 5 minutes after each injection with the ZENEO® injector at Day 1, after each MRI and at each follow-up visit (Day 3 and Day 6) of each treatment period.
  By using Visual Analogic Scale (VAS)

OTHER OUTCOMES:
Safety Outcomes and Evaluation | At Day +8 after the last injection with the ZENEO® injector.
  Occurrence of Adverse Events (AEs)/Device Deficiency

CONTACTS AND LOCATIONS:
Overall Officials: Maxime LUU, MD, PhD, Principal Investigator — CHU DIJON Bourgogne - Hôpital François Mitterrand
Locations (1):
- CHU DIJON Bourgogne - Hôpital François Mitterrand, Dijon, France

IPD SHARING:
Plan to Share IPD: No